CLINICAL TRIAL: NCT00022737
Title: A Children's Oncology Group Pilot Study for the Treatment of Very High Risk Acute Lymphoblastic Leukemia in Children and Adolescents (Imatinib (STI571, GLEEVEC) NSC#716051)
Brief Title: Combination Chemotherapy With or Without Peripheral Stem Cell Transplant in Treating Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01862; NCI-2012-01862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068859; COG-AALL0031; AALL0031 (Other: Children's Oncology Group); AALL0031 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2012-11

CONDITIONS: Childhood Acute Lymphoblastic Leukemia in Remission; Recurrent Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Asparaginase; palmitoyl-L-asparaginase; Cyclophosphamide; Cyclosporine; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; Etoposide; Ifosfamide; indolepropanol phosphate; Imatinib Mesylate; Leucovorin; Mercaptopurine; Methotrexate; merphos; pegaspargase; Vincristine; Transplantation; Peripheral Blood Stem Cell Transplantation; Cord Blood Stem Cell Transplantation; Radiotherapy; Radiation

ARMS (1):
- Arm I (Experimental): See Design Details.
  Interventions: Biological: filgrastim; Drug: asparaginase; Drug: cyclophosphamide; Drug: cyclosporine; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: etoposide; Drug: ifosfamide; Drug: imatinib mesylate; Drug: leucovorin calcium; Drug: mercaptopurine tablet; Drug: methotrexate; Drug: pegaspargase; Drug: vincristine sulfate; Procedure: allogeneic bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Procedure: umbilical cord blood transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Drug: asparaginase — Given IM
  Other Names: ASNase; Colaspase; Crasnitin; Elspar; L-ASP
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: cyclosporine — Given IV
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: cytarabine — Given IT and IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
Drug: dexamethasone — Given orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Drug: leucovorin calcium — Given IV or orally
  Other Names: CF; CFR; LV
Drug: mercaptopurine tablet — Given orally
  Other Names: 6-mercaptopurine; 6-MP; Leukerin; MP
Drug: methotrexate — Given IT, IV, and orally
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: pegaspargase — Given IM
  Other Names: L-asparaginase with polyethylene glycol; Oncaspar; PEG-ASP; PEG-L-asparaginase
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Procedure: allogeneic bone marrow transplantation — Undergo allogeneic bone marrow, peripheral blood stem cell, or umbilical cord blood transplantation
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic bone marrow, peripheral blood stem cell, or umbilical cord blood transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: umbilical cord blood transplantation — Undergo allogeneic bone marrow, peripheral blood stem cell, or umbilical cord blood transplantation
  Other Names: cord blood transplantation; transplantation, umbilical cord blood; UCB transplantation
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
This phase II trial is studying how well combination chemotherapy with or without donor peripheral stem cell transplant works in treating children with acute lymphoblastic leukemia. Giving combination chemotherapy before a donor peripheral stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of treatment with intensified chemotherapy, in terms of toxicity and patient accrual, in children with very high-risk acute lymphoblastic leukemia.

II. Determine the feasibility and efficacy of following intensified chemotherapy with allogeneic hematopoietic stem cell transplantation in patients with HLA-matched related donors.

III. Determine the toxicity of imatinib mesylate in combination with intensified chemotherapy in Philadelphia chromosome-positive patients.

IV. Determine the event-free survival of patients treated with this regimen. V. Determine whether minimal residual disease (MDR) after induction therapy and prior to intensification therapy can predict relapse in these patients.

VI. Determine whether MDR after intensification is prognostically significant. VII. Determine whether gene expression patterns predict disease recurrence or response to imatinib mesylate.

OUTLINE: This is a multicenter study. This is also a dose-escalation study of imatinib mesylate in Philadelphia chromosome-positive (Ph+) patients. Patients are stratified according to Philadelphia chromosome (Ph) status (Ph-positive vs Ph-negative or indeterminate), hypodiploidy (yes vs no), MLL translocation (11q23) AND slow early response to prior induction therapy (yes vs no), and failed prior induction therapy (yes vs no).

Cohorts of 8-12 Ph+ patients receive escalating doses of imatinib mesylate, according to the guidelines for each treatment block of this study, until the maximum tolerated dose (MTD) for each treatment combination is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 35 patients are treated at the MTD.

CONSOLIDATION BLOCK 1: Patients receive etoposide IV over 1 hour followed by ifosfamide IV over 1.5 hours on days 1-5. Patients also receive methotrexate intrathecally on day 1 and filgrastim (G-CSF) subcutaneously (SC) on days 6-15 or until blood counts recover. Patients with CNS 2/3 at diagnosis also receive intrathecal triple therapy comprising methotrexate, hydrocortisone, and cytarabine (ITT) on days 8 and 15. Ph+ patients in cohorts 3, 4, and 5 receive oral imatinib mesylate on days 1-21. Within 4 days of starting consolidation therapy, patients with biopsy-proven testicular leukemia undergo radiotherapy daily for 12 days.

CONSOLIDATION BLOCK 2: Patients receive high-dose methotrexate IV over 24 hours and ITT on day 1 followed by high-dose cytarabine IV over 3 hours, every 12 hours on days 2 and 3. Patients also receive leucovorin calcium IV or orally every 6 hours for 3 doses beginning on day 2, and G-CSF SC on days 4-13 or until blood counts recover. Ph+ patients in cohorts 2, 3, 4, and 5 receive oral imatinib mesylate as in consolidation block 1. Patients undergoing allogeneic hematopoietic stem cell transplantation (HSCT) proceed to preparative chemotherapy. All other patients proceed to reinduction block 1.

REINDUCTION BLOCK 1: Patients receive vincristine IV on days 1, 8, and 15; daunorubicin IV on days 1 and 2; cyclophosphamide IV over 30 minutes, every 12 hours on days 3 and 4; pegaspargase intramuscularly (IM) on day 4; and ITT on days 1 and 15. Patients also receive oral dexamethasone twice daily on days 1-7 and 15-21 and G-CSF SC on days 5-14 or until blood counts recover. Ph+ patients in cohorts 2, 4, and 5 receive imatinib mesylate as in consolidation block 1.

INTENSIFICATION BLOCK 1: Patients receive high-dose methotrexate IV over 24 hours on days 1 and 15 and ITT on days 1 and 22. Patients also receive leucovorin calcium IV or orally every 6 hours for 3 doses beginning on days 2 and 16. Patients receive etoposide IV over 2 hours followed by cyclophosphamide IV over 30 minutes on days 22-24; G-CSF SC on days 27-36 or until blood counts recover; high-dose cytarabine IV over 3 hours, every 12 hours on days 43 and 44; and asparaginase IM on day 44. Ph+ patients in cohorts 1 and 4 receive oral imatinib mesylate on days 43-63, and patients in cohort 5 receive oral imatinib mesylate on days 1-56.

REINDUCTION BLOCK 2: Patients receive vincristine, daunorubicin, cyclophosphamide, pegaspargase, dexamethasone, and G-CSF as in reinduction block 1. Patients also receive ITT on days 1 and 15. Ph+ patients receive imatinib mesylate as in reinduction block 1.

INTENSIFICATION BLOCK 2: Patients receive methotrexate, leucovorin calcium, etoposide, cyclophosphamide, filgrastim, cytarabine, and asparaginase as in intensification block 1. Ph+ patients receive imatinib mesylate as in intensification block 1.

MAINTENANCE 1: Patients receive high-dose methotrexate IV and leucovorin calcium as in consolidation block 2. Patients also receive ITT and vincristine IV on days 1 and 29; oral dexamethasone twice daily on days 1-5 and 29-33; oral methotrexate on days 8, 15, and 22; oral mercaptopurine on days 8-28; etoposide IV over 2 hours followed by cyclophosphamide IV over 30 minutes on days 29-33; and G-CSF SC on days 34-43. Ph+ patients in cohorts 1-4 receive oral imatinib mesylate on days 29-49 and patients in cohort 5 receive oral imatinib mesylate on days 1-56. Treatment repeats every 8 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE 2: Patients receive vincristine and dexamethasone as in maintenance 1. Beginning on day 1, patients undergo cranial radiotherapy once daily, 5 days a week, for approximately 2 weeks. Patients also receive oral methotrexate on days 8, 15, 22, 29, 36, 43, and 50 and oral mercaptopurine on days 11-56. Ph+ patients in cohorts 1-4 receive oral imatinib mesylate on days 1-21 and 29-49, and patients in cohort 5 receive oral imatinib mesylate on days 1-56.

MAINTENANCE 3: Patients receive vincristine and dexamethasone as in maintenance 2. Patients also receive oral methotrexate on days 1, 8, 15, 22, 29, 36, 43, and 50; and oral mercaptopurine on days 1-56. Ph+ patients receive imatinib mesylate as in maintenance 2. Treatment repeats every 8 weeks for 7 courses (12 courses total in maintenance 1, 2, and 3) in the absence of disease progression or unacceptable toxicity.

Patients may undergo allogeneic HSCT after consolidation block 2 if there is an available HLA-DR matched or HLA-A or -B matched or 1 antigen mismatched relative donor.

Patients with CNS leukemia undergo cranial radiotherapy 3 times daily on days -10 to -8. All patients undergo radiotherapy twice daily on days -7 to -5 and receive etoposide IV on day -4 and cyclophosphamide IV on days -3 and -2. Patients undergo allogeneic bone marrow, peripheral blood stem cell, or umbilical cord blood transplantation on day 0. Patients receive cyclosporine IV beginning on day -1 and continuing every 12 hours, switching to oral administration when possible, until day 60 and tapering thereafter. Patients also receive methotrexate on days 1, 3, and 6. Beginning 16-24 weeks after transplantation, Ph+ patients receive oral imatinib mesylate once daily for 24 weeks.

Patients are followed every 4-8 weeks for 1 year, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter. Patients undergoing HSCT are followed weekly for the first year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia
* Received prior front-line therapy on a Pediatric Oncology Group (POG),Children's Cancer Group (CCG), or Central Oncology Group (COG) study
* Received induction therapy comprising vincristine, asparaginase, prednisone/dexamethasone, and daunorubicin as in CCG, POG, or COG protocols
* M1 or M2 bone marrow status after front-line induction therapy and presenting with at least 1of the following:

  * Philadelphia chromosome positive (Ph+) with t(9;22)(q34;q11) by cytogenetics or fluorescence in situ hybridization
  * bcr-abl fusion transcript by reverse transcription polymerase chain reaction
  * Hypodiploid with less than 44 chromosomes and/or DNA index less than0.81
  * MLL translocation (11q23) by cytogenetics and a slow early response (SER) to induction therapy, defined as at least 5% blasts at day 15 of induction and/or at least .1% minimal residual disease (MRD) after induction therapy
* Failed to achieve remission after front-line induction therapy

  * M3 bone marrow status (greater than 25% blasts) after induction therapy
  * M2 bone marrow status (5-25% blasts) or at least 1% MRD after induction therapy and M2 or M3or at least 1% MRD after consolidation therapy (CCG studies) or extended induction therapy (POG or COG studies)
* See Disease Characteristics
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* See Disease Characteristics
* See Disease Characteristics
* No concurrent prophylactic cranial radiotherapy

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2002-10; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Feasibility, in terms of patient accrual | Up to 1.75 years
  As a target goal, we wish to enroll at least 80% of the potential available patients. The accrual duration for this pilot study will be based on accruing adequate numbers to complete the dose escalation study in the Ph+ subset. The planned study accrual duration should be approximately 1.75 years.
Feasibility, in terms of incidence of adverse events graded according to NCI CTC v 2.0 | Up to 7 years
  The use of imatinib as given in combination with other agents in a particular cohort will be considered feasible initially if 5 or more of the first 6 evaluable patients complete the phase(s) without evidence of grade 3 or 4 targeted toxicities.

SECONDARY OUTCOMES:
Event-free survival | Up to 7 years
  Estimated with 90% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Schultz, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States

REFERENCES:
- [Derived] Tasian SK, Peters C. Targeted therapy or transplantation for paediatric ABL-class Ph-like acute lymphocytic leukaemia? Lancet Haematol. 2020 Dec;7(12):e858-e859. doi: 10.1016/S2352-3026(20)30369-0. No abstract available. PMID 33242441